CLINICAL TRIAL: NCT06872268
Title: THERAPEUTIC PHOTOGRAPHY AND EXPRESSIVE WRITING: AN EXPLORATORY SEQUENTIAL MIXED-METHODS FEASIBILITY STUDY OF PATIENTS WITH MARFAN SYNDROME
Brief Title: APPLICATION OF THERAPEUTIC PHOTOGRAPHY AND EXPRESSIVE WRITING IN THE MANAGEMENT OF PATIENTS WITH MARFAN SYNDROME
Acronym: FOTOTEMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Policlinico S. Donato (Other)
Responsible Party: Principal Investigator, Alessandro Pini, Referent, IRCCS Policlinico S. Donato
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: FOTOTEMA
Record Dates: First submitted 2025-01-17; First posted 2025-03-12 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Marfan Syndrome
Keywords: therapeutic photography; expressive writing activities; Marfan syndrome; standard practice; mixed methods study
MeSH Terms: conditions — Marfan Syndrome

STUDY DESIGN:
Intervention Model Description: mixed-methods sequential exploratory study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention group (Experimental): Subjects with Marfan syndrome in follow-up at Cardiovascular Genetic Center, IRCCS Policlinico San Donato
  Interventions: Behavioral: Therapeutic photography and expressive writing; Behavioral: Expressive writing

INTERVENTIONS:
Behavioral: Therapeutic photography and expressive writing — Therapeutic photography, unlike phototherapy, consists of a set of photography-based activities that are initiated independently as part of an organised group or project, but in which no formal therapy is taking place within a psychotherapeutic setting. This approach, too, can be used as a routine practice in treatment pathways. The subject deepens his or her self-awareness to improve the sense of being: images become a way to express oneself, to communicate what one is unable to verbalize. Therapeutic photography can be done independently and individually, or in the presence of other professionals (nurses, sociologists, teachers, facilitators, psychologists) who accompany the individual to the understanding and production of the activity.
Behavioral: Expressive writing — Expressive writing is a technique that helps to understand and manage one's experiences and emotional tensions, contributes to mental and physical well-being, decreased stress, improved relationships, and the strengthening of the immune system.

SUMMARY:
This study explores the efficacy of therapeutic photography and expressive writing as interventions in routine practice for patients with Marfan syndrome.

DETAILED DESCRIPTION:
The objective of the study is to assess the feasibility of including structured therapeutic photography and expressive writing activities in routine practice as an adjunct to standard treatment for patients with Marfan syndrome in a national Reference Centre for Rare Diseases. This will include measuring the adherence rate to the programme and evaluating the subjective experience of the patients involved.

ELIGIBILITY:
Inclusion Criteria:

Subjects with Marfan syndrome referred to the Cardiovascular genetic center in IRCCS Policlinico San Donato;

- Signed informed consent.

Exclusion Criteria:

* Patients who are currently going through a period of severe medical or psychological instability reported in medical history.
* Subjects who are unable to provide informed consent due to cognitive, language, or other limitations that prevent full understanding of the purpose and nature of the study.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2024-04-02 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Efficacy of therapeutic photography in clinical practice | 18 months
  This approach will be assessed through semi-structured interviews and thematic analysis of photographs generated by participants to deepen their personal experience of living with a rare disease
Efficacy of expressive writing in clinical practice | 18 months
  This approach will be assessed through semi-structured interviews and thematic analysis texts generated by participants to deepen their personal experience of living with a rare disease

SECONDARY OUTCOMES:
Impact of therapeutic photography | 18 months
  Detect and compare the impact of therapeutic photography activities on patients and their perception of its effect in their care. This approach will be assessed through semi-structured interviews and thematic analysis of photographs generated by participants to deepen their personal experience of living with a rare disease
Impact of expressive writing | 18 months
  Detect and compare the impact of expressive writing activities on patients and their perception of its effect in their care. This approach will be assessed through semi-structured interviews and thematic analysis of texte written by participants to deepen their personal experience of living with a rare disease
Pre- and post-activity effects of therapeutic photography: patients' perspective | 18 months
  Psychological General Well-Being Index (PGWBI) questionnaire will be applied for the evaluation of this outcome
Pre- and post-activity effects of expressive writing: patients' perspective | 18 months
  Exploring patients' perceptions of attractiveness, efficiency, clarity, reliability, stimulation and originality of the program through standardized evaluations as a measure of proximity of feasibility.
Qualitative analysis | 18 months
  Exploring the experience of the patients involved with qualitative analysis of interviews, texts and photographs.

CONTACTS AND LOCATIONS:
Overall Officials: Nathasha Samali UDUGAMPOLAGE, MSN, Principal Investigator — IRCCS Policlinico S. Donato
Locations (1):
- IRCCS Policlinico San Donato, San Donato Milanese, Italy, Italy

IPD SHARING:
Plan to Share IPD: No
IPD will be shared after study closure.

REFERENCES:
- [Background] Panetta M, Bianchetti A, Udugampolage NS, Taurino J, Caruso R, Pini A, Callus E. Discussing psychological and psychotherapeutic support for patients with Marfan syndrome (MFS) and their family: an example of a structured program in Italy. Front Psychol. 2023 Jun 15;14:1176692. doi: 10.3389/fpsyg.2023.1176692. eCollection 2023. No abstract available. PMID 37397303
- [Background] Gibson, Neil. (2017). Therapeutic photography: enhancing patient communication. Journal of Kidney Care. 2. 46-47. 10.12968/jokc.2017.2.1.46.